CLINICAL TRIAL: NCT02353208
Title: The Effect of Sham Feeding on Small Bowel Transit Time in Patients Undergoing Capsule Endoscopy: a Prospective Randomized Trial
Brief Title: The Effect of Sham Feeding on Small Bowel Transit Time in Patients Undergoing Capsule Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Robert Enns, Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H14-03443
Record Dates: First submitted 2015-01-12; First posted 2015-02-02 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Slow Transit

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Feeding of Bacon Bits (Active Comparator): In addition to the standard procedure, subjects will be asked to perform sham feeding on two occasions: 1) Immediately after having swallowed the capsule and 2) One hour after having swallowed the capsule.
  Sham feeding will be performed as follows: The patients will be asked to chew 10 times on a piece of bacon over a period of 30 seconds, prior to spitting saliva and bacon into a container. This will be repeated 10 times at one minute intervals.
  The patient will then complete the capsule study as per the standard procedure.
  Bacon bits will be a commercially available produce which has been deemed safe for sale in Canada.
  Interventions: Other: Sham Feeding of Bacon Bits
- Placebo (Placebo Comparator): The control group will not chew bacon bits while undergoing capsule endoscopy.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Sham Feeding of Bacon Bits — Bacon bits will be a commercially available produce which has been deemed safe for sale in Canada.
  Other Names: Bacon bits
  Arms: Sham Feeding of Bacon Bits
Other: Placebo — Participants will not be asked to chew bacon bits
  Other Names: Control
  Arms: Placebo

SUMMARY:
Capsule endoscopy is a non-invasive way to examine the small bowel, but its yield is limited by the battery life. In 20% of cases, the recording stops before the entire length of small bowel is examined. Capsule transit speed is dependent on bowel motility. When we eat, the brain sends signal to the bowel to speed up motility. In this study the investigators wish to determine if chewing bacon (sham feeding) can trick the brain to speed up bowel motility and improve the rate of complete small bowel examination.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blinded controlled trial.

Subjects ages 19 years and older referred for capsule endoscopy (CE) at the GI Clinic, St. Paul's Hospital will be invited to participate in the study. We will be recruiting 122 subjects and will randomize them into 2 groups: control group and treatment group. Control subjects will undergo the standard capsule endoscopy procedure. Subjects in Treatment group will undergo sham feeding in addition to the standard capsule endoscopy procedure. Both control and treatment subjects in this study will be required to swallow a capsule (the size of a large pill) named Given Imaging SB3® Capsule.

The investigator and the video reader will be blinded (single-blinded study). Times will be recorded at: first gastric image, first duodenal image and first cecal image.

The diagnostic yield for controls and subjects will be calculated. The clarity of the images will be graded according to the ICCE 2005 consensus regarding bowel preparation and prokinetics in capsule endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients, 19 years or older referred to St. Paul's Hospital for capsule endoscopy

Exclusion Criteria:

* In-patients will be excluded
* Patients who have been taking taken medications that affect your bowel movement in the five days prior to the procedure
* Patients who are vegetarian or have dietary restrictions that do not allow bacon/pork products.
* Patients, who have proven or suspected obstruction of the bowel.
* Patients, who have had prior small bowel and/or stomach surgery.
* Patients who have a known and/or have a history suggestive of a swallowing disorder
* Patients with complicated diabetes diabetes with associated complications (bleeding in eyes, kidney disease, or numbness/tingling in hands/feet)
* Patient who have thyroid problem that is not being treated (for example, hypothyroid but not taking supplement)
* Patients who are pregnant, prisoners or an institutionalized individuals
* Patients whose capsule camera is placed using a traditional scope (instead of swallowing the capsule camera)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-01; Primary Completion 2016-11-16 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Small bowel transit time | 5 hours
  To investigate whether sham feeding using bacon shortens small bowel transit time (SBTT)

SECONDARY OUTCOMES:
Gastric transit time | 1 hour
  To investigate whether sham feeding shortens gastric transit time (GTT)
Diagnostic yield of capsule endoscopy | 5 hours
  To investigate whether sham feeding alters clarity of the capsule endoscopy images.
Completion examination rate | 8 hours
  To investigate whether sham feeding using bacon increases the completion examination rate (CER)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Enns, M.D., Principal Investigator — University of British Columbia
Locations (1):
- GI Clinic, St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] ASGE Technology Committee; Wang A, Banerjee S, Barth BA, Bhat YM, Chauhan S, Gottlieb KT, Konda V, Maple JT, Murad F, Pfau PR, Pleskow DK, Siddiqui UD, Tokar JL, Rodriguez SA. Wireless capsule endoscopy. Gastrointest Endosc. 2013 Dec;78(6):805-815. doi: 10.1016/j.gie.2013.06.026. Epub 2013 Oct 8. PMID 24119509
- [Background] Pasha SF, Leighton JA, Das A, Harrison ME, Decker GA, Fleischer DE, Sharma VK. Double-balloon enteroscopy and capsule endoscopy have comparable diagnostic yield in small-bowel disease: a meta-analysis. Clin Gastroenterol Hepatol. 2008 Jun;6(6):671-6. doi: 10.1016/j.cgh.2008.01.005. Epub 2008 Mar 20. PMID 18356113
- [Background] Iaquinto G, Fornasarig M, Quaia M, Giardullo N, D'Onofrio V, Iaquinto S, Di Bella S, Cannizzaro R. Capsule endoscopy is useful and safe for small-bowel surveillance in familial adenomatous polyposis. Gastrointest Endosc. 2008 Jan;67(1):61-7. doi: 10.1016/j.gie.2007.07.048. PMID 18155426
- [Background] Marmo R, Rotondano G, Piscopo R, Bianco MA, Cipolletta L. Meta-analysis: capsule enteroscopy vs. conventional modalities in diagnosis of small bowel diseases. Aliment Pharmacol Ther. 2005 Oct 1;22(7):595-604. doi: 10.1111/j.1365-2036.2005.02625.x. PMID 16181299
- [Background] Schulmann K, Hollerbach S, Kraus K, Willert J, Vogel T, Moslein G, Pox C, Reiser M, Reinacher-Schick A, Schmiegel W. Feasibility and diagnostic utility of video capsule endoscopy for the detection of small bowel polyps in patients with hereditary polyposis syndromes. Am J Gastroenterol. 2005 Jan;100(1):27-37. doi: 10.1111/j.1572-0241.2005.40102.x. PMID 15654777
- [Background] Triester SL, Leighton JA, Leontiadis GI, Fleischer DE, Hara AK, Heigh RI, Shiff AD, Sharma VK. A meta-analysis of the yield of capsule endoscopy compared to other diagnostic modalities in patients with obscure gastrointestinal bleeding. Am J Gastroenterol. 2005 Nov;100(11):2407-18. doi: 10.1111/j.1572-0241.2005.00274.x. PMID 16279893
- [Background] Caddy GR, Moran L, Chong AK, Miller AM, Taylor AC, Desmond PV. The effect of erythromycin on video capsule endoscopy intestinal-transit time. Gastrointest Endosc. 2006 Feb;63(2):262-6. doi: 10.1016/j.gie.2005.07.043. PMID 16427932
- [Background] Postgate A, Tekkis P, Patterson N, Fitzpatrick A, Bassett P, Fraser C. Are bowel purgatives and prokinetics useful for small-bowel capsule endoscopy? A prospective randomized controlled study. Gastrointest Endosc. 2009 May;69(6):1120-8. doi: 10.1016/j.gie.2008.06.044. Epub 2009 Jan 18. PMID 19152909
- [Background] Rondonotti E, Herrerias JM, Pennazio M, Caunedo A, Mascarenhas-Saraiva M, de Franchis R. Complications, limitations, and failures of capsule endoscopy: a review of 733 cases. Gastrointest Endosc. 2005 Nov;62(5):712-6; quiz 752, 754. doi: 10.1016/j.gie.2005.05.002. PMID 16246685
- [Background] Westerhof J, Weersma RK, Koornstra JJ. Risk factors for incomplete small-bowel capsule endoscopy. Gastrointest Endosc. 2009 Jan;69(1):74-80. doi: 10.1016/j.gie.2008.04.034. Epub 2008 Aug 8. PMID 18691709
- [Background] Aparicio JR, Martinez J, Casellas JA. Right lateral position does not affect gastric transit times of video capsule endoscopy: a prospective study. Gastrointest Endosc. 2009 Jan;69(1):34-7. doi: 10.1016/j.gie.2008.03.1111. Epub 2008 Jul 11. PMID 18620344
- [Background] Liao Z, Li F, Li ZS. Right lateral position improves complete examination rate of capsule endoscope: a prospective randomized, controlled trial. Endoscopy. 2008 Jun;40(6):483-7. doi: 10.1055/s-2007-995689. PMID 18556803
- [Background] Koulaouzidis A, Giannakou A, Yung DE, Dabos KJ, Plevris JN. Do prokinetics influence the completion rate in small-bowel capsule endoscopy? A systematic review and meta-analysis. Curr Med Res Opin. 2013 Sep;29(9):1171-85. doi: 10.1185/03007995.2013.818532. Epub 2013 Jul 11. PMID 23790243
- [Background] Power ML, Schulkin J. Anticipatory physiological regulation in feeding biology: cephalic phase responses. Appetite. 2008 Mar-May;50(2-3):194-206. doi: 10.1016/j.appet.2007.10.006. Epub 2007 Oct 24. PMID 18045735
- [Background] Defilippi C, Valenzuela JE. Sham feeding disrupts the interdigestive motility complex in man. Scand J Gastroenterol. 1981;16(8):977-9. doi: 10.3109/00365528109181014. PMID 7336138
- [Background] Stern RM, Crawford HE, Stewart WR, Vasey MW, Koch KL. Sham feeding. Cephalic-vagal influences on gastric myoelectric activity. Dig Dis Sci. 1989 Apr;34(4):521-7. doi: 10.1007/BF01536327. PMID 2702882
- [Background] Katschinski M, Dahmen G, Reinshagen M, Beglinger C, Koop H, Nustede R, Adler G. Cephalic stimulation of gastrointestinal secretory and motor responses in humans. Gastroenterology. 1992 Aug;103(2):383-91. doi: 10.1016/0016-5085(92)90825-j. PMID 1634057
- [Background] Brin VB, Tsabolova ZT. [The effect of calcitonin on the mechanisms of urine formation and sodium excretion in normotensive and spontaneously hypertensive rats]. Biull Eksp Biol Med. 1991 Feb;111(2):118-20. Russian. PMID 1854946
- [Background] Ou G, Svarta S, Chan C, Galorport C, Qian H, Enns R. The effect of chewing gum on small-bowel transit time in capsule endoscopy: a prospective, randomized trial. Gastrointest Endosc. 2014 Apr;79(4):630-6. doi: 10.1016/j.gie.2013.08.038. Epub 2013 Oct 7. PMID 24112594
- [Background] Feldman M, Richardson CT. Role of thought, sight, smell, and taste of food in the cephalic phase of gastric acid secretion in humans. Gastroenterology. 1986 Feb;90(2):428-33. doi: 10.1016/0016-5085(86)90943-1. PMID 3940915
- [Background] Abdallah L, Chabert M, Louis-Sylvestre J. Cephalic phase responses to sweet taste. Am J Clin Nutr. 1997 Mar;65(3):737-43. doi: 10.1093/ajcn/65.3.737. PMID 9062523
- [Background] Wicks D, Wright J, Rayment P, Spiller R. Impact of bitter taste on gastric motility. Eur J Gastroenterol Hepatol. 2005 Sep;17(9):961-5. doi: 10.1097/00042737-200509000-00012. PMID 16093874
- [Background] Schiller LR, Feldman M, Richardson CT. Effect of sham feeding on gastric emptying. Gastroenterology. 1980 Jun;78(6):1472-5. PMID 7372066
- [Background] Soffer EE, Adrian TE. Effect of meal composition and sham feeding on duodenojejunal motility in humans. Dig Dis Sci. 1992 Jul;37(7):1009-14. doi: 10.1007/BF01300279. PMID 1618049
- [Background] Powley TL, Berthoud HR. Diet and cephalic phase insulin responses. Am J Clin Nutr. 1985 Nov;42(5 Suppl):991-1002. doi: 10.1093/ajcn/42.5.991. PMID 3933326
- [Background] Teff KL, Devine J, Engelman K. Sweet taste: effect on cephalic phase insulin release in men. Physiol Behav. 1995 Jun;57(6):1089-95. doi: 10.1016/0031-9384(94)00373-d. PMID 7652029
- [Background] de Franchis R, Avgerinos A, Barkin J, Cave D, Filoche B; ICCE. ICCE consensus for bowel preparation and prokinetics. Endoscopy. 2005 Oct;37(10):1040-5. doi: 10.1055/s-2005-870327. No abstract available. PMID 16189787